CLINICAL TRIAL: NCT04228666
Title: A Clinical Trial to Determine the Safety and Efficacy of Hope Biosciences Autologous Mesenchymal Stem Cell Therapy (HB-adMSCs) for the Treatment of Alzheimer's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to COVID 19 Pandemic
Sponsor: Hope Biosciences LLC (Industry)
Collaborators: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBALZ01
Record Dates: First submitted 2020-01-03; First posted 2020-01-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; stem cells; adipose derived mesenchymal stem cells
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB-adMSCs (Experimental): HB-adMSCs are autologous, adipose-derived mesenchymal stem cells. Four intravenous infusions will be administered on weeks 0, 2, 6, and 8 at a dose of 2 x 10^8 total HB-adMSC cells.
  Interventions: Biological: HB-adMSCs

INTERVENTIONS:
Biological: HB-adMSCs — Four IV infusions of autologous adipose-derived mesenchymal stem cells. Baseline laboratory data will be collected prior to first infusion; follow-up data will be compared against baseline according to the following schedule: safety laboratory tests follow-up on weeks 4, 8, 13, 26, and 52; inflammation and amyloid markers follow-up on weeks 13 and 52; MMSE and ADCS-ADL follow-up on weeks 13, 19, 26, 33, 40, 46 and 52; Altoida NMI follow-up will occur weekly from week 0 to week 52; CDR follow-up will occur weeks 4, 10, 13, 19, 26, 33, 40, 46 and 52; C-SSRS follow-up will occur on weeks 4, 10, 26, and 52; Amyloid PET imaging follow-up occurs week 26 and 52;

SUMMARY:
Hope Biosciences is conducting a research study of an investigational product called autologous adipose-derived mesenchymal stem cells (abbreviated as HB-adMSCs) as a possible treatment for Alzheimer's disease (AD). The study purpose is to evaluate the safety profile of four IV infusions of HB-adMSCs in subjects with clinical diagnosis of AD.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, non-randomized study in subjects with Alzheimer's disease. 24 patients will be enrolled for the study. The overall objective of this study is to evaluate the safety profile of four IV infusions of autologous adipose-derived mesenchymal stem cells (HB-adMSCs) in subjects with clinical diagnosis of AD. The primary endpoint of this study is to measure the number and frequency of adverse event(s) and/or severe adverse event(s) throughout the study duration. The second endpoint of this study is to evaluate the ability of HB-adMSCs to alter AD-related inflammation via measuring levels of Tumor Necrosis Factor alpha (TNF-a), Interleukin-1 (IL-1), Interleukin-6 (IL-6), C-Reactive Protein (CRP), and markers associated with amyloid deposition, Amyloid beta 40 and Amyloid beta 42. Subjects will also be assessed for cognitive deficits measured by changes from baseline values using Mini Mental Status Examination (MMSE), Alzheimer's disease Cooperative Study Activities of Daily Living (ADCS-ADL), Alzheimer's disease Related Quality of Life (ADRQL), Altoida Neuro Motor Index (NMI) for Digital Biomarkers, and Clinical Dementia Rating Questionnaire (CDR).

ELIGIBILITY:
Inclusion Criteria:

1. Men, and women of non-childbearing potential, 50-85 years of age inclusively, with a diagnosis of early stage's (preclinical/mild cognitive impairment) Probable Alzheimer's Disease according to the 2011 NIA-AA criteria.

   * Non-childbearing potential for women is defined as postmenopausal [last natural menses greater than 24 months; in women under age 55, menopausal status will be documented with serum follicle stimulating hormone (FSH) test] or undergone a documented bilateral tubal ligation or hysterectomy.
   * Male participants who are sexually active with a woman of childbearing potential must agree to use condoms during the trial unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of intrauterine device (IUD), male or female condom and diaphragm.
2. Informed consent signed by the subject
3. Documented Amyloid PET Scan (images and report) positive to amyloid plaques deposits on the brain.
4. If the patient is under any treatment, should have been on a stable dose for at least 30 days prior to signing the informed consent form and there is no intention to modify the dose over the course of the study. (NOTE: Cholinesterase inhibitors (AChEI) (donepezil, galantamine, or rivastigmine) may not be initiated, discontinued or modified after study initiation for the 12-months control period).

Exclusion Criteria:

1. Hospitalization or change of chronic concomitant medication within one month prior to screening.
2. Clinically significant or unstable disease that may interfere with outcome evaluations, including but not limited to:

   * Respiratory Insufficiency
   * Poorly managed hypertension (systolic >160 mm Hg and/or diastolic >95 mm Hg) or hypotension (systolic <90 mm Hg and/or diastolic <60 mm Hg); or
   * Bradycardia (<50 beats/min.) or tachycardia (>100 beats/min.). Otherwise healthy subjects with borderline bradycardia may be discussed with the medical monitor to determine eligibility.
   * Renal insufficiency, defined as eGFR <40 mL/min based on the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula, https://www.mdcalc.com/ckd-epi-equations-glomerular-filtration-rate-gfr
   * Heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within 3 months before screening). If a subject has a history of heart disease of questionable clinical significance, the medical monitor may be contacted to discuss eligibility.
3. Records of PET Scan negative to Amyloid plaques deposition in the brain.
4. Suspected or known drug or alcohol abuse, i.e. more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day.
5. Acute intercurrent infections such as Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), Human Immunodeficiency Virus (HIV) or Syphilis.
6. Contraindications for PET scanning, including implanted metallic devices (e.g. non-MRI-safe cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces.
7. Is unable or unwilling to comply with protocol follow-up requirements.
8. Enrollment in another investigational study or intake of investigational drug within the previous 30 days.
9. Any condition, which in the opinion of the investigator or the sponsor makes the patient unsuitable for inclusion.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Glucose | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of glucose in the blood (mg/dL)
Calcium | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of calcium in the blood (mg/dL)
Albumin | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of albumin in the blood (g/dL)
Total Protein | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of protein in the blood (g/dL)
Sodium | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of sodium in the blood (mol/L)
Total carbon dioxide | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of carbon dioxide in the blood (mmol/L)
Potassium | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of potassium in the blood (mmol/L)
Chloride | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of chloride in the blood (mmol/L)
BUN | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of BUN in the blood (mg/dL)
Creatinine | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of creatinine in the blood (mg/dL)
Alkaline phosphatase | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of alkaline phosphatase in the blood (IU/L)
Alanine aminotransferase | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of alanine aminotransferase in the blood (IU/L)
Aspartate aminotransferase | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of aspartate aminotransferase in the blood (IU/L)
Total Bilirubin | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of bilirubin in the blood (mg/dL)
White blood cell | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of white blood cells in the blood (x 10^3/uL)
Red blood cell | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of red blood cells in the blood (x 10^6/uL)
Hemoglobin | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of hemoglobin in the blood (g/dL)
Hematocrit | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of hematocrit in the blood (%)
Mean corpuscular volume | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of mean corpuscular volume in the blood (fL)
Mean corpuscular hemoglobin | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of mean corpuscular hemoglobin in the blood (pg)
Mean corpuscular hemoglobin concentration | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of level of hemoglobin concentration in the blood (g/dL)
Red cell distribution width | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of distribution width in the blood (%)
Neutrophils | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of neutrophils in the blood (%)
Lymphs | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of lymphocytes in the blood (%)
Monocytes | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of monocytes in the blood (%)
Eos | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of eosinophils in the blood (%)
Basophils | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of basophils in the blood (%)
Absolute neutrophils | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of absolute neutrophils in the blood (x 10^3/uL)
Absolute lymphs | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of absolute lymphocytes in the blood (x 10^3/uL)
Absolute monocytes | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of absolute monocytes in the blood (x 10^3/uL)
Absolute Eos | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of absolute eosinophils in the blood (x 10^3/uL)
Absolute Basos | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of absolute basophils in the blood (x 10^3/uL)
Immature granulocytes | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of granulocytes in the blood (%)
Absolute Immature granulocytes | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of absolute immature granulocytes in the blood (x 10^3/uL)
Platelets | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of platelets in the blood (x 10^3/uL)
Prothrombin time | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of time for blood to coagulate (seconds)
INR | Screening, change from screening at week 0, week 4, week 8, week 13, week 26, week 52.
  clinical lab evaluation of international normalized ratio of blood coagulation (no unit)

SECONDARY OUTCOMES:
Tumor necrosis factor-alpha | week 0, change from baseline at week 13, change from baseline at week 52
  measure level of TNFa in blood (pg/ml)
Interleukin-1 | week 0, change from baseline at week 13, change from baseline at week 52
  measure of IL-1 in the blood (pg/ml)
Interleukin-6 | week 0, change from baseline at week 13, change from baseline at week 52
  measure of IL-6 in the blood (pg/ml)
C-reactive protein | week 0, change from baseline at week 13, change from baseline at week 52
  measure of CRP in the blood (mg/L)
Amyloid beta 40 | week 0, change from baseline at week 13, change from baseline at week 52
  measure of AB40 in the blood (pg/ml)
Amyloid beta 42 | week 0, change from baseline at week 13, change from baseline at week 52
  measure of AB42 in the blood (pg/ml)
Volumetric changes in hippocampus, ventriculus, and whole brain | screening, week 26 and 52
  volume change from screening
Mini Mental Status Exam | week 0, change from baseline at week 4, 10, 13, 19, 26, 33, 40, 46, and 52
  Change from baseline score; scores from 0 to 30, lower score indicates more severe dementia
Alzheimer's disease Cooperative Study Activities of Daily Living | week 0, change from baseline at week 4, 10, 13, 19, 26, 33, 40, 46, and 52
  Change from baseline score; scores from 0 to 53, lower score indicates greater functional impairment
Quality of Life Enjoyment and Satisfaction Questionnaire | week 0, change from baseline at week 4, 10, 13, 19, 26, 33, 40, 46, and 52
  Change from baseline score; total score range is 14 to 70, higher scores indicate more enjoyment and satisfaction with life
Altoida Neuro Motor Index | week 0, change from baseline at week 4, 10, 13, 19, 26, 33, 40, 46, and 52
  Change from baseline score; score ranges from 0 to 100, higher score indicates less impairment
Clinical Dementia Rating Questionnaire | week 0, change from baseline at week 4, 10, 13, 19, 26, 33, 40, 46, and 52
  Change from baseline score; scores range fro 0 to 3, higher scores indicates more severe impairment

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Clinical Trial Network
Locations (1):
- Clinical Trial Network, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No